CLINICAL TRIAL: NCT02686957
Title: Risk Factors of Fistula Recurrence and Pregnancy Outcomes Following Fistula Repair in Guinea
Brief Title: Recurrence and Pregnancy Post-repair of Obstetric Fistula in Guinea
Status: Completed | Type: Observational
Sponsor: Centre National de Formation et de Recherche en Sante Rurale (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Other Study IDs: ITM948/14
Record Dates: First submitted 2016-02-12; First posted 2016-02-22 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women closed: This cohort will include women who underwent repair for obstetric fistula at three fistula repair hospitals in Guinea and who had a closed fistula at hospital discharge.
  no intervention will be done.

SUMMARY:
Obstetric fistula, also called vaginal fistula, is a serious medical condition which affects women in low income countries. Despite the strengthening of research on fistula, there is little data on the follow-up after fistula repair.

The objective of this study is to analyse the factors associated with the recurrence of fistula and the outcomes of pregnancy following fistula repair in Guinea. It will target women who got a closed fistula at discharge after repair in 2012/2015 at three fistula repair sites supported by the Fistula Care Project in Guinea (Kissidougou Prefectoral Hospital, Labé Regional Hospital and Jean Paul II Hospital of Conakry).

The outcomes of interest are fistula recurrence and pregnancy. The predictors of interest will include patient characteristics, fistula characteristics, the context of repair and the context of reintegration.

Participants giving an informed consent after a home visit by the Fistula Counsellors who managed women during surgery will be interview at enrolment and every six month from inclusion. The study duration is estimated at 48 months (January 2012 to March 2016) including the retrospective part.

A sample size of 364 women will estimate the recurrence of fistula with a plus/minus 2% margin of error (width of confidence interval is 4%) and 95% confidence interval and is sufficient to estimate the rate of pregnancy with a two-sided 95% confidence interval and 10% precision.

The cumulative incidence rate of fistula recurrence will be calculated using Kaplan-Meier methods and the risk factor analysis will be performed using adjusted cox regression.

For the outcomes of pregnancy, Pearson's Chi Square (χ2) will be used to compare proportions of pregnancy outcomes between potential predictors and logistic regression models will be used and associations will be reported as risk ratios with 95% confidence intervals.

Analysis will be done using STATA version 13 (STATA Corporation, College Station, TX, USA) with a level of significance set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible, study participants must meet the following criteria:

* Had a fistula closed at discharge, as measured by a dye test (this include women dry and those with residual incontinence);
* Willing and able to provide written informed consent (assent for minors);
* Had a urinary or recto-vaginal fistula;
* Agree to participate in follow-up visits (every six months) from consent date and for the duration of the study;
* Agree to stay in Guinea for the duration of the study.

Exclusion Criteria:

Potential participants meeting any of the following criteria will not be enrolled in the study:

* Refusal to give free and informed consent;
* Surgery done outside the study sites;
* Incomplete medical records;
* Incontinence unrelated to urinary or recto-vaginal fistula.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of women who underwent repair for obstetric fistula in three fistula repair hospitals in Guinea from 1 January 2012 to 30 June 2015.
Sampling Method: Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Recurrence of fistula | 2012-2015, up to 8 months
  Recurrence of fistula is defined as a "continuous and uncontrolled leakage of urine" in a woman up to 48 months after hospital discharge.

SECONDARY OUTCOMES:
Pregnancy | 2012-2016, up to 48 months
  Pregnancy is defined by a positive pregnancy test (medical records) or a self-reporting confirmed by at least two witnesses in a woman up to 48 months after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DELAMOU, MD, PhDcand, Principal Investigator — Centre National de Formation et de Recherche en Sante Rurale
Locations (1):
- Centre National de Formation et de Recherche en Sante Rurale, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: No
Such data will not be public unless requested and after prior authorization of the Guinean National Ethics Committee for Health Research.

REFERENCES:
- [Derived] Delamou A, Delvaux T, Beavogui AH, Leveque A, Zhang WH, De Brouwere V. A descriptive longitudinal study protocol: recurrence and pregnancy post-repair of obstetric fistula in Guinea. BMC Pregnancy Childbirth. 2016 Oct 10;16(1):299. doi: 10.1186/s12884-016-1101-y. PMID 27724918